CLINICAL TRIAL: NCT04753060
Title: Hair Cycle Modulation To Promote Human Wound Healing
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study suspended temporarily due to coronavirus pandemic.
Sponsor: University of Hull (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Matthew Hardman, Chief Investigator, University of Hull
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: RS105
Record Dates: First submitted 2021-02-02; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Wounds
Keywords: Wound; Hair Follicle
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waxing (Active Comparator): Waxing of patients donor site who are undergoing a skingraft procedure, prior to surgery taking place.
  Interventions: Procedure: Waxing
- Standard care (No Intervention): Standard wound preparation

INTERVENTIONS:
Procedure: Waxing — Donor sites of patients skin grafts are waxed prior to surgery for donor harvesting.
  Arms: Waxing

SUMMARY:
Chronic wounds represent a huge burden to both patients and the National Health Service (NHS), with over 200,000 sufferers in the UK alone. Based on current conservative estimates the NHS spends £2.3 - £3.1 billion pounds every year treating these patients.

This study aims to reduce this shared burden, preliminary data from our research group using animal models has demonstrated variable ability of hair follicles to heal wounds based upon their stage within their growth cycle. This currently proposed study therefore aims to perform a simple novel intervention on patients prior to their elective surgery in an effort to replicate the substantial healing abilities noted in the animal models.

Under normal circumstances, a patient's operative site is shaved prior to the surgery for hygiene and visual simplicity. The aim of this study is to wax 50% of the patient's operative site prior to their surgery, the other half will be shaved on the day of surgery as per normal surgical protocol. Based on known data this waxing technique will cycle the hair follicles into their growth phase at the time of surgery. The growth phase of hair follicles corresponds with an increased ability to heal due to recruitment of a patients own stem cells. This study therefore aims to take advantage of the patient's own stem cell population. The 50% waxing and 50% shaving method upon each patients donor site allows us to directly compare the influence of these two methods directly on a patient-by-patient basis.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing skin graft surgery
* Patient is 18 years of age or older.
* Written and informed consent provided.

Exclusion Criteria:

* Participants that have been enrolled in a clinical trial within the last 3 months that would affect their ability to heal or influence hair cycle.
* Specific hair-linked diseases, e.g. alopecia areata. (Not including androgenetic alopecia)
* Lack of capacity to consent
* Lymphedema
* Malnutrition
* Collagen disorders
* Patients requiring grafts smaller than 5cm x 5cm
* Patients requiring grafts wider than 10cm
* Immunomodulation drugs
* Patients will be excluded mid study if they develop an infection that prevents biopsy retrieval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Photograph Assessment | 7 days post-surgery
  Digital assessment of healing outcome from clinical wound photographs using novel scale (1-10). Higher score is representative of a better outcome.
Photograph Assessment | 14 days post-surgery
  Digital assessment of healing outcome from clinical wound photographs using novel scale (1-10). Higher score is representative of a better outcome.
Photograph Assessment | 3 months post-surgery
  Digital assessment of healing outcome from clinical wound photographs using novel scale (1-10). Higher score is representative of a better outcome.

SECONDARY OUTCOMES:
Post Operative Infection incidence | 7 days post surgery
  Clinical assessment reports a presence or absence of infection
Post Operative Infection incidence | 14 days post surgery
  Clinical assessment reports a presence or absence of infection
Post Operative Infection incidence | 3 months post surgery
  Clinical assessment reports a presence or absence of infection
Changes To Patient Microbiome (Next-Generation Sequencing) | 0, 7, 14 days and 3 months.
  Changes to skin microbiome as compared to day 0 using next-generation sequencing.
Histological Wound Healing Score | Day 0
  H&E stained histological sections will be used to quantify healing using a study-specific scale (1-10). Higher score is representative of an improved outcome.
Histological Wound Healing Score | 7 days post surgery
  H&E stained histological sections will be used to quantify healing using a study-specific scale (1-10). Higher score is representative of an improved outcome.
Histological Wound Healing Score | 14 days post surgery
  H&E stained histological sections will be used to quantify healing using a study-specific scale (1-10). Higher score is representative of an improved outcome.
Histological Wound Healing Score | 3 months post surgery
  H&E stained histological sections will be used to quantify healing using a study-specific scale (1-10). Higher score is representative of an improved outcome.
Identification of Hair Cycle State via Histology | Day 0
  Tissue biopsies will be analysed histologically to identify the presence of anagen and telogen hair follicles.
Identification of Hair Cycle State via Histology | 7 days post surgery
  Tissue biopsies will be analysed histologically to identify the presence of anagen and telogen hair follicles.
Identification of Hair Cycle State via Histology | 14 days post surgery
  Tissue biopsies will be analysed histologically to identify the presence of anagen and telogen hair follicles.

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Hill Hospital, Hull, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared but non-identifiable results will be published in an appropriate journal.